CLINICAL TRIAL: NCT06125574
Title: The Effects of Regular OMT on Stress Levels and Cognitive Function in OMS-I Students at Touro COM-NY Harlem
Brief Title: Investigating the Effects of Osteopathic Manipulative Treatment on Stress Management in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Touro College and University System (Other)
Responsible Party: Principal Investigator, Mikhail Volokitin, MD, DO., Assistant Professor, The Touro College and University System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18777
Record Dates: First submitted 2023-11-04; First posted 2023-11-09 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Stress, Job; Student Burnout; Stress, Physiological; Stress, Psychological
Keywords: Osteopathic Manipulative Medicine; Osteopathic Manipulative Treatment; OMM; OMT; Cortisol; Medical Student Stress; Cognitive Function
MeSH Terms: conditions — Occupational Stress; Burnout, Psychological; Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Other: Osteopathic Manipulative Medicine
- Control (No Intervention)

INTERVENTIONS:
Other: Osteopathic Manipulative Medicine — Individuals in the experimental cohort will undergo a systematic osteopathic manipulative treatment protocol encompassing paraspinal inhibition, rib raising, and condylar decompression techniques.
  Arms: Treatment

SUMMARY:
The goal of this clinical trial is to evaluate stress biomarkers, subjective stress levels, and cognitive function in medical students. The main question[s] it aims to answer are:

Does regular osteopathic manipulative treatment affect stress in medical students? Does regular osteopathic manipulative treatment affect cognitive function in medical students?

Participants will be split into two groups, control and treatment, and undergo a designated protocol for six weeks. The treatment protocol will include weekly sessions of three OMT techniques: paraspinal inhibition, rib raising, and condylar decompression. Concurrently, participants' salivary cortisol levels will be collected weekly and analyzed using an Invitrogen ELISA Immunoassay Kit. Additionally, cognitive function will be assessed weekly via Lumosity, while stress levels are gauged using the College Student Stress Scale (CSSS) survey.

Researchers will compare one cohort of medical students who receive weekly OMT and another cohort of medical students who have weekly check-ins without OMT to see if OMT can affect changes in stress biomarkers, subjective stress scales, and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* First-year medical students
* Not currently receiving osteopathic manipulative treatment (OMT)

Exclusion Criteria:

* Pregnant
* History of spinal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Weekly Cortisol Level | Weekly, over the course of 8 week study
  Salivary Cortisol as measured in an ELISA Immunoassay
College Student Subjective Stress Survey (CSSS) Numerical Score | Weekly, over the course of 8 week study
  Numerical Score collected from the College Student Subjective Stress Survey, a 10-item survey investigating occurrence of stressors over the course of a week, with each item being rated from 1 (Never) to 5 (Very Often). A lower score reflects lower perceived stress while a higher score reflects higher perceived stress.
LPI | Weekly, over the course of 8 week study
  Learning Performance Index Metric from Lumosity

CONTACTS AND LOCATIONS:
Locations (1):
- Touro College of Osteopathic Medicine - Harlem, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bath M, Owens J. Physiology, Viscerosomatic Reflexes. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559218/ PMID 32644644
- [Background] Degenhardt BF, Darmani NA, Johnson JC, Towns LC, Rhodes DC, Trinh C, McClanahan B, DiMarzo V. Role of osteopathic manipulative treatment in altering pain biomarkers: a pilot study. J Am Osteopath Assoc. 2007 Sep;107(9):387-400. PMID 17908831
- [Background] Feldt RC. Development of a brief measure of college stress: the college student stress scale. Psychol Rep. 2008 Jun;102(3):855-60. doi: 10.2466/pr0.102.3.855-860. PMID 18763455
- [Background] Licciardone JC, Kearns CM, Hodge LM, Bergamini MV. Associations of cytokine concentrations with key osteopathic lesions and clinical outcomes in patients with nonspecific chronic low back pain: results from the OSTEOPATHIC Trial. J Am Osteopath Assoc. 2012 Sep;112(9):596-605. doi: 10.7556/jaoa.2012.112.9.596. PMID 22984233
- [Background] Licciardone JC, Schultz MJ, Amen B. Osteopathic Manipulation in the Management of Chronic Pain: Current Perspectives. J Pain Res. 2020 Jul 20;13:1839-1847. doi: 10.2147/JPR.S183170. eCollection 2020. PMID 32765058
- [Background] Lee BK, Glass TA, McAtee MJ, Wand GS, Bandeen-Roche K, Bolla KI, Schwartz BS. Associations of salivary cortisol with cognitive function in the Baltimore memory study. Arch Gen Psychiatry. 2007 Jul;64(7):810-8. doi: 10.1001/archpsyc.64.7.810. PMID 17606815
- [Background] Saeed SMU, Anwar SM, Khalid H, Majid M, Bagci AU. EEG based Classification of Long-term Stress Using Psychological Labeling. Sensors (Basel). 2020 Mar 29;20(7):1886. doi: 10.3390/s20071886. PMID 32235295
- [Background] Schoorlemmer RM, Peeters GM, van Schoor NM, Lips P. Relationships between cortisol level, mortality and chronic diseases in older persons. Clin Endocrinol (Oxf). 2009 Dec;71(6):779-86. doi: 10.1111/j.1365-2265.2009.03552.x. Epub 2009 Feb 18. PMID 19226268
- [Background] Shute, V. J., Ventura, M., & Ke, F. (2015). The power of play: The effects of portal 2 and lumosity on cognitive and noncognitive skills. Computers & Education, 80, 58-67.